CLINICAL TRIAL: NCT06779227
Title: Implementation Ond Evaluation of Hospital-to-Home Transitional Care Intervention in Patients with Chronic Heart Failure
Brief Title: Implementation and Evaluation of Hospital-to-Home Transitional Care Intervention in Patients with Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhi-fen Feng (Other)
Responsible Party: Sponsor-Investigator, Zhi-fen Feng, Associate Professor, School of Nursing and Health, Henan University, Henan University
Organization: Henan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUSOM2021-289
Record Dates: First submitted 2024-12-30; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): The control group received routine care.
- Intervention group (Experimental): The intervention group received a transitional care intervention mainly focused on the transitional care model (TCM).
  Interventions: Behavioral: Hospital family transitional nursing intervention

INTERVENTIONS:
Behavioral: Hospital family transitional nursing intervention — The intervention group received a transitional care intervention mainly focused on the transitional care model (TCM).
  Arms: Intervention group

SUMMARY:
This study lasted for a total of three months. The purpose is to build a hospital-family transitional nursing intervention program for patients with chronic heart failure, and to explore the effectiveness of the program on the self-management of patients with chronic heart failure, in order to provide certain empirical research for the clinical intervention of transitional nursing for patients with chronic heart failure. If you have any questions or difficulties, you can withdraw from this study at any time, which will not affect your treatment and nursing. The purpose of this study is to improve your self-care level and prevent your re-admission. It will not harm your physical and mental health and will not have a negative impact on the relationship between patients and nursing. You participate in this study and The personal data in the study is confidential, and any public report on the results of this study will not disclose your personal identity.

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of the New York Heart Association (NYHA) for CHF, and the heart function level is II to III;
* Age ≥18 years old;
* The condition is stable and meets the standard of being discharged from the hospital;
* Clear consciousness, no communication barriers, able to understand and fill in the questionnaire correctly;
* Informed consent and voluntary participation in this study.

Exclusion Criteria:

* Patients with hepato-renal disfunction, sequelae of stroke, dementia;
* Patients with a history of mental disorders or already having mental disorders, critically ill patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Self-efficacy management indicators | Baseline, one month, three months
  The measurement tool adopts the Chronic Disease Self-Efficacy Questionnaire compiled by Stanford University in the United States.The scoring consists of two dimensions: symptom management and disease-commonality management. The self-efficacy score for symptom management is calculated by averaging items 1, 2, 3, and 4 (if two or more items are missing or omitted, the variable is considered missing). A higher score indicates greater self-efficacy in symptom management. The self-efficacy score for disease-commonality management is obtained by averaging items 5 and 6. The score ranges from 1 to 5, a higher score indicates higher self-efficacy in disease-commonality management.

SECONDARY OUTCOMES:
Self-care indicators | Baseline, one month, three months
  In this study, the Chinese version of the self-care ability scale for elderly, translated by Guo , was used. The scale demonstrates good reliability and validity, with a Cronbach's α coefficient of 0.82, a test-retest reliability of 0.82, and a content validity index of 0.94. The scale consists of 17 items and is applicable to all older adults. Scoring on the scale ranges from "completely disagree" to "completely agree," with scores ranging from 1 to 5. Higher scores indicate a higher self-care ability in older adults.
Disease-related indicators | Baseline, one month, three months
  Disease-related indicators are the indicators of frequent examination of patients with heart failure in the hospital: The blood test index adopts NT-proBNP as a measurement indicator, which is an independent risk factor for the death and re-admission of patients with heart failure. Due to structure and metabolism, NT-pro BNP has the advantages of long half-life (120min), high blood concentration, low individual variability rate, good in vitro stability, not limited by specimen collection conditions and the influence of specimen type (plasma or serum). NT-pro BNP testing on patients can help assess long-term risks. Repeated determination will provide more prognostic information for patients.
Transitional nursing evaluation indicators | Baseline, one month, three months
  This study adopts the Care Transitions Measure (CTM-15) developed by American scholar COLEMAN in 2002. This scale is a self-assessment scale that evaluates transitional care from the patient's perspective, including information transmission ( 6 items), patient participation (3 entries), management preparation (4 entries), nursing plan (2 entries) 4 dimensions, a total of 15 entries. The results show that the total scale Cronbach's α coefficient is 0.93, and the content validity index is 0.99, which has good credibility. The scores of each item: "very disagree", "disagree", "agree" and "very agree" are 1~4 points respectively, and the final score is converted to 0~100 points. The higher the score, indicating that the research subjects are satisfied with the transitional nursing services.

OTHER OUTCOMES:
Re-hospitalisation indicators | Baseline, one month, three months
  The study mainly measures the re-hospitalisation of the study subjects and whether the re-hospitalisation rate of the two groups has changed. By counting the re-admission of the study subjects, the re-admission rate of the two groups is calculated, which is mainly collected through the combination of the hospital's HIS system inquiry and asking patients or family members. HIS's scoring adopts the method of multi-dimensional evaluation. Each dimension contains multiple items, and each item has a corresponding scoring standard. The scoring generally adopts the five-level method, from 0 to 4 points, indicating no impact, mild impact, moderate impact, severe impact and very serious impact respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nursing and Health, School of Nursing and Health, Henan University, Kaifeng, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng ZF, Liu Y, Salvador JT, Ala MB, Nery MAC, Huang XY, Zhang L, Liu S. Implementation and evaluation of hospital-to-home transitional care intervention in patients with chronic heart failure. BMC Nurs. 2025 Jul 1;24(1):717. doi: 10.1186/s12912-025-03447-5. PMID 40597265